







Version 2.0 20-Feb-19 Centre: PIN: REC Number: IRAS ID: 256260

## PARENTAL CONSENT FORM

## This consent form is for parents/carers of participants aged 12-15

## Online PTSD treatment for Young People and their Carers (OPTYC): Case Series Dr Patrick Smith

| | | Please initial box | |
|---|---|---|---|
| 1. | I have been consulted about my child's particle opportunity to ask questions about the stutheir taking part in this research. | | |
| 2. | I understand that my child's participation is voluntary and that I can request that they are withdrawn from the study at any time without giving any reason, and without their medical care or legal rights being affected. | | |
| 3. | I understand that relevant data collected during the study about my child, may be looked at by individuals from King's College London, from regulatory authorities or from the NHS Trust, where it is relevant to their taking part in this research. I give permission for these individuals to have access to my child's records. | | |
| 4. | I understand that the information collected about my child will be used to support other research in the future, and may be shared anonymously with other researchers. | | |
| 5. | I understand that my child's relevant confidential information will be disclosed to appropriate professionals, including their GP, if a clinical or research worker on the study becomes concerned about my child's, or someone else's safety. | | |
| 6. | I agree to my child's General Practitioner being informed of their participation in the study and being involved in the study, including any necessary exchange of information about me between my GP and the research team. | | |
| 7. | I understand that the information held and maintained by South London and Maudsley NHS Foundation Trust may be used to help contact my child or provide information about their health status. | | |
| 8. | I agree for my child to take part in the above study. | | |
| our | Name Relationship to child | Date | Signature |
| lame of Person taking consent | | Date | Signature |